CLINICAL TRIAL: NCT05044715
Title: Effectiveness of Compassion Focused Therapy (CFT) Adapted to a Group Format: Outcomes and Mechanisms of Change
Brief Title: Effectiveness of Compassion Focused Therapy (CFT)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The prevalence of CFT at the counseling center and university made it difficult during recruitment of subjects to find participants without exposure to CFT to be used as a treatment-as-usual control.
Sponsor: Brigham Young University (Other)
Responsible Party: Principal Investigator, Gary Burlingame, Professor/Department Chair, Clinical Psychology, Brigham Young University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB2020-220
Record Dates: First submitted 2021-08-06; First posted 2021-09-16 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Compassion; Self-Criticism; Shame; Guilt
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Members will be randomized to treatment-as-usual (TAU) CAPS groups or CFT groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (Experimental): Participants in this arm will receive treatment as usual (TAU) as an intervention.
  Interventions: Behavioral: Treatment as Usual
- Compassion-Focused Therapy (Experimental): Participants in this arm will be enrolled in a CFT group intervention.
  Interventions: Behavioral: Compassion-Focused Therapy (CFT)

INTERVENTIONS:
Behavioral: Treatment as Usual — Treatment as usual-TAU groups include:
  1. Mood Groups - General Process Groups
  2. Anxiety Groups - Cognitive Behavioral Therapy
  3. Body Image and Eating Concerns Groups
  4. Reconciling Faith and Sexuality Groups
  Arms: Treatment as Usual
Behavioral: Compassion-Focused Therapy (CFT) — The CFT protocol assumes that participants have no prior experience with meditation, mindfulness, and self-compassion and teaches principles of each as well as skills such as guided meditations.
  Arms: Compassion-Focused Therapy

SUMMARY:
The proposed study is a randomized controlled trial (RCT) that takes place at Brigham Young University's (BYU) Counseling and Psychological Services (CAPS). The proposed study follows from the CAPS open trial which led to revisions of the compassion-focused therapy (CFT) protocol authored by Paul Gilbert. In essence, the study is taking existing evidence-based group treatments offered at CAPS, and comparing patient outcomes in a systematic manner. The investigators intend to replicate the improvement rates observed in the open trial with the revised CFT protocol and ascertain if outcomes are comparable to members who receive treatment-as-usual-TAU CAPS groups and those receiving CFT.

Hypotheses:

1. Group members attending a 12-session CFT group will have higher levels of compassion and self-reassurance as well as lower levels of self-criticism (and self-hate), fears of compassion, shame, and psychiatric distress when compared to members attending the parallel TAU groups.
2. Amount of change in compassion, self-reassurance, self-criticism (and self-hate), fears of compassion, and shame will be comparable for CFT measures authored by Dr. Gilbert as measures developed by independent compassion researchers.
3. There will be comparable levels of change in general psychiatric distress, as measured by the Outcome Questionnaire -45 (OQ-45), in members attending CFT and TAU groups. However, there will be greater change in members attending CFT groups on measures of compassion.
4. CFT will lead to lower levels of internalized shame through the mechanisms of fear reduction and increases in the 3 flows of compassion.

DETAILED DESCRIPTION:
Compassion-based interventions (CBIs) have become popular in the last ~30 years, either as standalone interventions or adjuncts to other treatments. Compassion focused therapy (CFT) is a CBI that was originally designed to be an adjunct to other interventions (e.g., individual psychotherapy). The focus on increasing compassion (especially self-compassion) grew out of the recognition that self-compassion has a strong positive relationship with well-being and a mirroring negative relationship with psychopathology (i.e., depression and anxiety). Indeed, six identified CBIs have been subjected to rigorous testing in RCTs, finding a medium effect on average (d = 0.55) across outcomes (e.g., depression, distress, well-being). CFT is "the most evaluated, and is the most appropriate for use in clinical populations" of all CBIs. CFT's evidence basis is expansive, prompting researchers to compose a review of its benefits for different populations and presenting problems (e.g., psychotic-spectrum disorders, people wanting to quit smoking). Researchers called for large-scale and high-quality trials having larger samples to further evaluate CFT. In particular, they call for this research to clarify equivocal results on important outcomes (i.e., some nonsignificant reductions of self-criticism). They also called for the inclusion of comparison groups stating that the next step was demonstrate that it produces comparable effects to other evidence-based interventions. A limitation noted by researchers was the existing CFT research includes a range of session length (i.e., as low as one and up to 16 weeks) and strategies (e.g., using cognitive restructuring, letter-writing, client-chosen practice with audio recordings) which varied widely between research groups. Furthermore, a portion of the evidence basis for CFT involves its combination with other third-wave psychotherapeutic interventions (i.e., acceptance and commitment therapy). Taken together, CFT has been adapted in multiple ways and its quality of evidence needs to be expanded, strengthening measurement and research designs as well as employing a standardized protocol that can be replicated with fidelity at multiple settings. The above limitations in existing CFT research prompted an open trial testing the effectiveness and feasibility of a standardized CFT protocol created by Paul Gilbert for group therapy at BYU's CAPS. The intent was to refine the CFT protocol so that it could be used in randomized trials, such as the one proposed in the present study. The production and empirical refinement of the CFT protocol by the BYU CAPS open trial directly addresses a serious problem in existing CFT trials that use incomparable treatment protocols. The investigators' CFT protocol was designed to be delivered in a group format. The investigators' BYU lab (http://cgrp.byu.edu) has a long tradition of making an empirical case for equivalence of group and individual treatments when delivered with fidelity. Indeed, three recent papers by the investigators provide compelling evidence for format equivalence using findings from both highly controlled randomized clinical trials and daily practice. Prior to the open trial, CFT had been delivered using a group treatment format, but its use with clinical populations is embryonic. Thus, the investigators' goal is to integrate CFT treatment as a group intervention targeting college counseling center clients to provide a rigorous empirical test of CFT theory. The investigators intend to do this by comparing CFT to treatment-as-usual groups for various presenting problems (e.g., depression and anxiety, eating disorders and sexual concerns) over the course of group treatment. Doing so will answer the call for higher-quality evidence and evaluate if (a) the theory-specified path of self-criticism to shame is present in treatment groups, and (b) this path can be mediated by CFT using the model.

Aims:

1. To assess the effects of CFT with a college counseling center population by measuring self-criticism (including self-reassurance and self-hate), compassion (i.e., for self, others, and from others), fears of compassion, shame, guilt and psychiatric distress to replicate the open trial outcomes.
2. To assess differences in effectiveness due to measurement source. In the open trial, investigators used measures created by Paul Gilbert (a founder of CFT) and those developed by independent researchers. This study replicates the process used in the open trial and the investigators do so again to ascertain if there is a measurement bias.
3. To assess the differential effectiveness of CFT groups compared to treatment-as-usual (TAU) groups run in Brigham Young University's (BYU) Counseling and Psychological Services (CAPS). CFT group protocols have been developed for clients presenting with: (a) general distress-mood disorders, (2) anxiety disorders, (3) eating disorders, and (4) challenges reconciling intersecting identities of faith and/or sexuality. CAPS currently offers evidence-based groups for each of these populations (e.g., general process, anxiety, eating, and intersecting identities, respectively). The investigators will compare members in groups that are randomly assigned to parallel CFT or TAU groups on compassion and general distress measures.
4. To assess the effect of mediation between reducing the fears of compassion, increases in compassion and the final outcome of reducing self-criticism and shame. This effect has been reported in the CFT literature; however, the previous analyses did not adequately report parameters (e.g., the unmediated effect) making interpretation incomplete.

ELIGIBILITY:
Inclusion Criteria:

* Struggles with issues of shame or self-criticism
* Have an Outcome Questionnaire (OQ-45) total score at or above 64 (i.e., denoting psychiatric distress in the clinical range)
* Are willing to commit to at least 4 sessions of group treatment
* Are willing to complete the OQ-45 and GQ (standardized CAPS measures) on a weekly basis
* Are willing to have group be their primary mode of treatment to ensure group will be the primary vehicle for change
* Are willing to complete the study measures

Exclusion Criteria

* Clients who do not meet criteria or decline to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Fears of Compassion Scale (FCS) | Pre-treatment (prior to first session, with measures cut off at session two)
  The FCS is a 38-item scale measuring fears of compassion on a five-point scale (0 = don't agree at all to 4 = completely agree). The FCS includes three scales, with higher scores indicating greater fears of compassion. Scales include: (1) expressing compassion for others (minimum score: 0; maximum score: 40), (2) responding to the expression of compassion from others (minimum score: 0; maximum score: 52), and (3) expressing kindness and compassion toward the self (minimum score: 0; maximum score: 60).
Fears of Compassion Scale (FCS) | Mid-treatment (between week six and week seven of intervention)
  The FCS is a 38-item scale measuring fears of compassion on a five-point scale (0 = don't agree at all to 4 = completely agree). The FCS includes three scales, with higher scores indicating greater fears of compassion. Scales include: (1) expressing compassion for others (minimum score: 0; maximum score: 40), (2) responding to the expression of compassion from others (minimum score: 0; maximum score: 52), and (3) expressing kindness and compassion toward the self (minimum score: 0; maximum score: 60).
Fears of Compassion Scale (FCS) | Post-treatment (within two weeks of the conclusion of the twelfth group session)
  The FCS is a 38-item scale measuring fears of compassion on a five-point scale (0 = don't agree at all to 4 = completely agree). The FCS includes three scales, with higher scores indicating greater fears of compassion. Scales include: (1) expressing compassion for others (minimum score: 0; maximum score: 40), (2) responding to the expression of compassion from others (minimum score: 0; maximum score: 52), and (3) expressing kindness and compassion toward the self (minimum score: 0; maximum score: 60).
Fears of Compassion Scale (FCS) | 90-day assessment (90 days after completion of intervention)
  The FCS is a 38-item scale measuring fears of compassion on a five-point scale (0 = don't agree at all to 4 = completely agree). The FCS includes three scales, with higher scores indicating greater fears of compassion. Scales include: (1) expressing compassion for others (minimum score: 0; maximum score: 40), (2) responding to the expression of compassion from others (minimum score: 0; maximum score: 52), and (3) expressing kindness and compassion toward the self (minimum score: 0; maximum score: 60).
Compassionate Engagement and Action Scales (CEAS) | Pre-treatment (prior to first session, with measures cut off at session two)
  The CEAS is a 39-item scale. The CEAS includes three scales, including compassion for self, compassion for others, and compassion from others. A total score can be calculated for each subscale (minimum score: 10; maximum score: 100), with higher scores indicating greater compassionate engagement and action. Furthermore, each scale is divided into two subscales: engagement and action. For each scale, subscale scores can be calculated for engagement (minimum score: 6; maximum score: 60) and action (minimum score: 4; maximum score: 40).
Compassionate Engagement and Action Scales (CEAS) | Mid-treatment (between week six and week seven of intervention)
  The CEAS is a 39-item scale. The CEAS includes three scales, including compassion for self, compassion for others, and compassion from others. A total score can be calculated for each subscale (minimum score: 10; maximum score: 100), with higher scores indicating greater compassionate engagement and action. Furthermore, each scale is divided into two subscales: engagement and action. For each scale, subscale scores can be calculated for engagement (minimum score: 6; maximum score: 60) and action (minimum score: 4; maximum score: 40).
Compassionate Engagement and Action Scales (CEAS) | Post-treatment (within two weeks of the conclusion of the twelfth group session)
  The CEAS is a 39-item scale. The CEAS includes three scales, including compassion for self, compassion for others, and compassion from others. A total score can be calculated for each subscale (minimum score: 10; maximum score: 100), with higher scores indicating greater compassionate engagement and action. Furthermore, each scale is divided into two subscales: engagement and action. For each scale, subscale scores can be calculated for engagement (minimum score: 6; maximum score: 60) and action (minimum score: 4; maximum score: 40).
Compassionate Engagement and Action Scales (CEAS) | 90-day assessment (90 days after completion of intervention)
  The CEAS is a 39-item scale. The CEAS includes three scales, including compassion for self, compassion for others, and compassion from others. A total score can be calculated for each subscale (minimum score: 10; maximum score: 100), with higher scores indicating greater compassionate engagement and action. Furthermore, each scale is divided into two subscales: engagement and action. For each scale, subscale scores can be calculated for engagement (minimum score: 6; maximum score: 60) and action (minimum score: 4; maximum score: 40).
Forms of Self Criticism and Self Reassuring Scale (FSCRS) | Pre-treatment (prior to first session, with measures cut off at session two)
  The FSCRS is a 22-item scale developed to measure people's critical and self-reassuring responses to setbacks or disappointments on a five-point scale (ranging from 0 = not at all like me to 4 = extremely like me). The FSCRS measures two forms of self-criticalness (i.e., inadequate self and hated self) and one form to self-reassure (i.e., reassure self). A score can be calculated for the inadequate self (minimum score: 0; maximum score: 36), hated self (minimum score: 0; maximum score: 20), and reassure self (minimum score: 0; maximum score: 32), with higher scores indicating a stronger inadequate self, hated self, and reassure self, respectively.
Forms of Self Criticism and Self Reassuring Scale (FSCRS) | Mid-treatment (between week six and week seven of intervention)
  The FSCRS is a 22-item scale developed to measure people's critical and self-reassuring responses to setbacks or disappointments on a five-point scale (ranging from 0 = not at all like me to 4 = extremely like me). The FSCRS measures two forms of self-criticalness (i.e., inadequate self and hated self) and one form to self-reassure (i.e., reassure self). A score can be calculated for the inadequate self (minimum score: 0; maximum score: 36), hated self (minimum score: 0; maximum score: 20), and reassure self (minimum score: 0; maximum score: 32), with higher scores indicating a stronger inadequate self, hated self, and reassure self, respectively.
Forms of Self Criticism and Self Reassuring Scale (FSCRS) | Post-treatment (within two weeks of the conclusion of the twelfth group session)
  The FSCRS is a 22-item scale developed to measure people's critical and self-reassuring responses to setbacks or disappointments on a five-point scale (ranging from 0 = not at all like me to 4 = extremely like me). The FSCRS measures two forms of self-criticalness (i.e., inadequate self and hated self) and one form to self-reassure (i.e., reassure self). A score can be calculated for the inadequate self (minimum score: 0; maximum score: 36), hated self (minimum score: 0; maximum score: 20), and reassure self (minimum score: 0; maximum score: 32), with higher scores indicating a stronger inadequate self, hated self, and reassure self, respectively.
Forms of Self Criticism and Self Reassuring Scale (FSCRS) | 90-day assessment (90 days after completion of intervention)
  The FSCRS is a 22-item scale developed to measure people's critical and self-reassuring responses to setbacks or disappointments on a five-point scale (ranging from 0 = not at all like me to 4 = extremely like me). The FSCRS measures two forms of self-criticalness (i.e., inadequate self and hated self) and one form to self-reassure (i.e., reassure self). A score can be calculated for the inadequate self (minimum score: 0; maximum score: 36), hated self (minimum score: 0; maximum score: 20), and reassure self (minimum score: 0; maximum score: 32), with higher scores indicating a stronger inadequate self, hated self, and reassure self, respectively.
Self-criticism and Rumination Scale (SCRS) | Pre-treatment (prior to first session, with measures cut off at session two)
  The SCRS is a 10-item scale developed to measure trait self-critical rumination on a four-point scale (ranging from 1 = not at all to 4 = very well). The SCRS utilizes a mean score (minimum score: 0; maximum score: 4). Higher scores indicate more self-critical rumination.
Self-criticism and Rumination Scale (SCRS) | Mid-treatment (between week six and week seven of intervention)
  The SCRS is a 10-item scale developed to measure trait self-critical rumination on a four-point scale (ranging from 1 = not at all to 4 = very well). The SCRS utilizes a mean score (minimum score: 0; maximum score: 4). Higher scores indicate more self-critical rumination.
Self-criticism and Rumination Scale (SCRS) | Post-treatment (within two weeks of the conclusion of the twelfth group session)
  The SCRS is a 10-item scale developed to measure trait self-critical rumination on a four-point scale (ranging from 1 = not at all to 4 = very well). The SCRS utilizes a mean score (minimum score: 0; maximum score: 4). Higher scores indicate more self-critical rumination.
Self-criticism and Rumination Scale (SCRS) | 90-day assessment (90 days after completion of intervention)
  The SCRS is a 10-item scale developed to measure trait self-critical rumination on a four-point scale (ranging from 1 = not at all to 4 = very well). The SCRS utilizes a mean score (minimum score: 0; maximum score: 4). Higher scores indicate more self-critical rumination.
External and Internal Shame Scale (EISS) | Pre-treatment (prior to first session, with measures cut off at session two)
  The EISS is an 8-item scale developed to assess shame that is directed at the individual from external ("People around me see me as not being up to their standards") and internal ("I am an unworthy person") sources on a five-point scale (0 = never to 4 = always). The EISS has an external shame subscale (minimum score: 0; maximum score: 16) and an internal shame subscale (minimum score: 0; maximum score: 16), with 4 items for each, and also has a total scale score (minimum score: 0; maximum score: 32). Higher scores indicate more shame.
External and Internal Shame Scale (EISS) | Mid-treatment (between week six and week seven of intervention)
  The EISS is an 8-item scale developed to assess shame that is directed at the individual from external ("People around me see me as not being up to their standards") and internal ("I am an unworthy person") sources on a five-point scale (0 = never to 4 = always). The EISS has an external shame subscale (minimum score: 0; maximum score: 16) and an internal shame subscale (minimum score: 0; maximum score: 16), with 4 items for each, and also has a total scale score (minimum score: 0; maximum score: 32). Higher scores indicate more shame.
External and Internal Shame Scale (EISS) | Post-treatment (within two weeks of the conclusion of the twelfth group session)
  The EISS is an 8-item scale developed to assess shame that is directed at the individual from external ("People around me see me as not being up to their standards") and internal ("I am an unworthy person") sources on a five-point scale (0 = never to 4 = always). The EISS has an external shame subscale (minimum score: 0; maximum score: 16) and an internal shame subscale (minimum score: 0; maximum score: 16), with 4 items for each, and also has a total scale score (minimum score: 0; maximum score: 32). Higher scores indicate more shame.
External and Internal Shame Scale (EISS) | 90-day assessment (90 days after completion of intervention)
  The EISS is an 8-item scale developed to assess shame that is directed at the individual from external ("People around me see me as not being up to their standards") and internal ("I am an unworthy person") sources on a five-point scale (0 = never to 4 = always). The EISS has an external shame subscale (minimum score: 0; maximum score: 16) and an internal shame subscale (minimum score: 0; maximum score: 16), with 4 items for each, and also has a total scale score (minimum score: 0; maximum score: 32). Higher scores indicate more shame.

SECONDARY OUTCOMES:
Outcome Questionnaire-45 (OQ-45) | Weekly (12 weeks)
  The OQ-45 is a 45-item scale that measures client psychiatric distress on interpersonal relations, symptom distress, and social role performance on a five-point scale (ranging from 0 = never to 4 = almost always) (minimum score: 0; maximum score: 180). Higher scores indicate greater distress.
Group Questionnaire (GQ) | Weekly (12 weeks)
  The GQ is a 30 item measure of the quality of therapeutic relationship in groups. It is measured on a 7-point Likert scale from 1 (not true at all) to 7 (very true). There are three subscales, each scored individually: positive bonding relationship (minimum score: 13; maximum score: 91), positive working relationship (minimum score: 8; maximum score: 56), and negative relationship (minimum score: 9; maximum score: 63). There is no total score. Higher scores on positive bonding indicate a strong alliance. Higher scores on positive work indicate that the member is experiencing the group as meeting their expectations for the changes they seek in group and that the group is working together to achieve mutually agreed upon goals. Higher scores on negative relationship could indicate alliance rupture with the leader, empathic failure with other members, or conflict in the group.
CFT knowledge and skill assessment (KSA) | Weekly (11 weeks)
  The KSA was developed by the investigators. It assesses CFT knowledge and CFT skills, and asks member to identify which CFT practices they are using and the frequency of use. The goal of this tool is to assess the degree to which the member remembers key information and is using CFT behavioral practices, which is assessed for each module except for module 12. The number of questions varies per week from 2 to 5 questions. The KSA is scored according to the percentage of questions that the participant got right (minimum score: 0; maximum score: 1).

CONTACTS AND LOCATIONS:
Overall Officials: Gary M Burlingame, PhD, Principal Investigator — Brigham Young University
Locations (1):
- Brigham Young University, Provo, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is likely that all collected IPD data will be used in future studies that support programmatic research in BYU CAPS and the investigators' continuing research on compassion therapy. Confidentiality will be maintained by using an assigned ID number.

REFERENCES:
- [Background] Baumeister D, Sedgwick O, Howes O, Peters E. Auditory verbal hallucinations and continuum models of psychosis: A systematic review of the healthy voice-hearer literature. Clin Psychol Rev. 2017 Feb;51:125-141. doi: 10.1016/j.cpr.2016.10.010. Epub 2016 Nov 1. PMID 27866082
- [Background] Beavan V. Towards a definition of "hearing voices": A phenomenological approach. Psychosis. 2011; 3(1): 63-73. doi:10.1080/17522431003615622
- [Background] Braehler C, Gumley A, Harper J, Wallace S, Norrie J, Gilbert P. Exploring change processes in compassion focused therapy in psychosis: results of a feasibility randomized controlled trial. Br J Clin Psychol. 2013 Jun;52(2):199-214. doi: 10.1111/bjc.12009. Epub 2012 Oct 24. PMID 24215148
- [Background] Burlingame GM, Gleave R, Erekson D, Nelson PL, Olsen J, Thayer S, Beecher M. Differential effectiveness of group, individual, and conjoint treatments: An archival analysis of OQ-45 change trajectories. Psychother Res. 2016 Sep;26(5):556-72. doi: 10.1080/10503307.2015.1044583. Epub 2015 Jul 14. PMID 26170048
- [Background] Burlingame GM, Seebeck JD, Janis RA, Whitcomb KE, Barkowski S, Rosendahl J, Strauss B. Outcome differences between individual and group formats when identical and nonidentical treatments, patients, and doses are compared: A 25-year meta-analytic perspective. Psychotherapy (Chic). 2016 Dec;53(4):446-461. doi: 10.1037/pst0000090. PMID 27918191
- [Background] Chandwick P, Lees S, Birchwood M. The revised Beliefs About Voices Questionnaire (BAVQ-R). Br J Psychiatry. 2000 Sep;177:229-32. doi: 10.1192/bjp.177.3.229. PMID 11040883
- [Background] Chapman CL, Burlingame GM, Gleave R, Rees F, Beecher M, Porter GS. Clinical prediction in group psychotherapy. Psychother Res. 2012;22(6):673-81. doi: 10.1080/10503307.2012.702512. Epub 2012 Jul 10. PMID 22775060
- [Background] Corstens D, Longden E, McCarthy-Jones S, Waddingham R, Thomas N. Emerging perspectives from the hearing voices movement: implications for research and practice. Schizophr Bull. 2014 Jul;40 Suppl 4(Suppl 4):S285-94. doi: 10.1093/schbul/sbu007. PMID 24936088
- [Background] Weng HY, Fox AS, Shackman AJ, Stodola DE, Caldwell JZ, Olson MC, Rogers GM, Davidson RJ. Compassion training alters altruism and neural responses to suffering. Psychol Sci. 2013 Jul 1;24(7):1171-80. doi: 10.1177/0956797612469537. Epub 2013 May 21. PMID 23696200
- [Background] Dillon J. The tale of an ordinary little girl. Psychosis. 2010; 2(1): 79-83. doi:10.1080/17522430903384305
- [Background] Hammersley P, Read J, Woodall S, Dillon J. Childhood Trauma and Psychosis: The Genie Is Out of the Bottle. Journal of Psychological Trauma. 2008; 6(2-3): 7-20. doi:10.1300/j513v06n02_02
- [Background] Gilbert P, Procter S. Compassionate mind training for people with high shame and self-criticism: Overview and pilot study of a group therapy approach. Clinical Psychology and Psychotherapy. 2006; 13(6): 353.
- [Background] Gilbert P, Clarke M, Hempel S, Miles JN, Irons C. Criticizing and reassuring oneself: An exploration of forms, styles and reasons in female students. Br J Clin Psychol. 2004 Mar;43(Pt 1):31-50. doi: 10.1348/014466504772812959. PMID 15005905
- [Background] Goss K, Allan S. The development and application of compassion-focused therapy for eating disorders (CFT-E). Br J Clin Psychol. 2014 Mar;53(1):62-77. doi: 10.1111/bjc.12039. PMID 24588762
- [Background] Hofmann SG, Grossman P, Hinton DE. Loving-kindness and compassion meditation: potential for psychological interventions. Clin Psychol Rev. 2011 Nov;31(7):1126-32. doi: 10.1016/j.cpr.2011.07.003. Epub 2011 Jul 26. PMID 21840289
- [Background] Horwood V, Allan S, Goss K, Gilbert P. The development of the Compassion Focused Therapy Therapist Competence Rating Scale. Psychol Psychother. 2020 Jun;93(2):387-407. doi: 10.1111/papt.12230. Epub 2019 Apr 25. PMID 31021509
- [Background] Kelly A, Zuroff D, Foa C, Gilbert P. Who benefits from training in self-compassionate self-regulation? A study of smoking reduction. Journal of Social and Clinical Psychology. 2009; 29: 727-755.
- [Background] Khoury B, Lecomte T, Gaudiano BA, Paquin K. Mindfulness interventions for psychosis: a meta-analysis. Schizophr Res. 2013 Oct;150(1):176-84. doi: 10.1016/j.schres.2013.07.055. Epub 2013 Aug 15. PMID 23954146
- [Background] Krogel J, Burlingame G, Chapman C, Renshaw T, Gleave R, Beecher M, Macnair-Semands R. The Group Questionnaire: a clinical and empirically derived measure of group relationship. Psychother Res. 2013;23(3):344-54. doi: 10.1080/10503307.2012.729868. Epub 2013 Feb 22. PMID 23432457
- [Background] Leary MR, Tate EB, Adams CE, Allen AB, Hancock J. Self-compassion and reactions to unpleasant self-relevant events: the implications of treating oneself kindly. J Pers Soc Psychol. 2007 May;92(5):887-904. doi: 10.1037/0022-3514.92.5.887. PMID 17484611
- [Background] MacBeth A, Gumley A. Exploring compassion: a meta-analysis of the association between self-compassion and psychopathology. Clin Psychol Rev. 2012 Aug;32(6):545-52. doi: 10.1016/j.cpr.2012.06.003. Epub 2012 Jun 23. PMID 22796446
- [Background] Neff KD. The development and validation of a scale to measure self-compassion. Self and Identity. 2003; 2: 223-250.
- [Background] Neff KD. Self-compassion: An alternative conceptualization of a healthy attitude toward oneself. Self and Identity. 2003; 2: 85-102.
- [Background] Neff KD, Vonk R. Self-compassion versus global self-esteem: two different ways of relating to oneself. J Pers. 2009 Feb;77(1):23-50. doi: 10.1111/j.1467-6494.2008.00537.x. Epub 2008 Nov 28. PMID 19076996
- [Background] Neff KD, Hsieh Y, Dejitterat K. Self-compassion, achievement goals and coping with academic failure. Self and Identity. 2005; 4: 263-287.
- [Background] Read J, Agar K, Argyle N, Aderhold V. Sexual and physical abuse during childhood and adulthood as predictors of hallucinations, delusions and thought disorder. Psychol Psychother. 2003 Mar;76(Pt 1):1-22. doi: 10.1348/14760830260569210. PMID 12689431
- [Background] Rockliff H, Gilbert P, McEwan K, Lightman S, Glover D. A pilot exploration of heart rate variability and salivary cortisol responses to compassion-focused imagery. Clinical Neuropsychiatry. 2008; 5, 132-139.
- [Background] Sapey B, Bullimore P. Listening to voice hearers. Journal of Social Work. 2013; 13(6): 616-632. doi:10.1177/1468017312475278
- [Background] Teasdale JD, Segal ZV, Williams JM, Ridgeway VA, Soulsby JM, Lau MA. Prevention of relapse/recurrence in major depression by mindfulness-based cognitive therapy. J Consult Clin Psychol. 2000 Aug;68(4):615-23. doi: 10.1037//0022-006x.68.4.615. PMID 10965637
- [Background] Thayer S, Burlingame, G. The validity of the Group Questionnaire: Construct clarity or construct drift? Group Dynamics: Theory, Research and Practice. 2014; 18(4): 318-332. http://dx.doi.org/10.1037/gdn0000015
- [Background] Tirch DD. Mindfulness as a context for the cultivation of compassion. International Journal of Cognitive Therapy. 2010; 3(2): 113-123.
- [Background] Vaughan S, Fowler D. The distress experienced by voice hearers is associated with the perceived relationship between the voice hearer and the voice. Br J Clin Psychol. 2004 Jun;43(Pt 2):143-153. doi: 10.1348/014466504323088024. PMID 15169615